CLINICAL TRIAL: NCT03808896
Title: Taipei City Hospital ZhongXing Branch, Emergency Department
Brief Title: TCHCCT-Zhong-Xing-Emergency-Department-airway-clincal (TTC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Hung,Tzu-Yao, Director of emergency department, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCHCCT-ZXERRP
Record Dates: First submitted 2018-12-23; First posted 2019-01-18 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Intubation;Difficult; Intubation Complication

STUDY DESIGN:
Intervention Model Description: Traditional intubation technique direct and video laryngoscope, bougie-assisted intubation, intubation with stylet assisted epiglottis lifting
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bougie-assisted intubation (Active Comparator): use bougie as guide, intubation with loading endotracheal tube under direct or video laryngoscopy
  Interventions: Device: bougie-assisted intubation
- intubation with epiglottic lifting (Active Comparator): Lifting of epiglottis with stylet-equipped endotracheal tube to assist intubation under direct or video laryngoscopy
  Interventions: Procedure: stylet-assisted epiglottic lifting
- Traditional intubation (No Intervention): intubation under direct or video laryngoscopy without epiglottis lifting nor bougie-assited

INTERVENTIONS:
Procedure: stylet-assisted epiglottic lifting — use stylet-equipped enodtracheal tube to lift the epiglottis and pass the endotracheal tube
  Arms: intubation with epiglottic lifting
Device: bougie-assisted intubation — use bougie as a introducer. Pass the bougie to the trachea and pass the tube via bougie guide.
  Other Names: bougie introducer
  Arms: bougie-assisted intubation

SUMMARY:
In the previous study on mannekin, the investigators found stylet-assisted lifting of epiglottis is an useful technique on difficult airway (Cormack-Lehane grade IIIa, IIIb) without increasing subjective difficulty. It has no expenses other than the routine intubation process. Recently, the studies have proved that the bougie-assisted laryngoscopy can improve first pass intubation rate in the emergency department. However, bougie is a disposable device and may increased medical expenditure. The investigators will evaluate the safety of bougie and epiglottic lifting technique, as well as the first pass and overall success rate of intubation comparing to traditional video laryngoscopy and direct laryngoscopy.

DETAILED DESCRIPTION:
A better strategy of managing Cormack-Lehane Grade III had been investigated by our previous study. The investigators' research results had been accepted and published by the journal BioMeidcal Central Anesthesiology. The investigators will be eager to do the further clinical trial to investigate the impact of this technique clinically. Besides, bougie assisted intubation is a effective, evidenced-proved intervention. The investigators will also like to find out the prognosis differences between these two techniques.

ELIGIBILITY:
Inclusion Criteria:

* all the patients present to the emergency department with airway emergency who need intubation

Exclusion Criteria:

* age below 18 year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2021-02-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
first pass success rate | through the intubation period, an average of 90 seconds
  first pass sucess rate
duration of intubation | through the intubation period, an average of 90 seconds

SECONDARY OUTCOMES:
Immediate complications direct related to intubation process | through the intubation period, an average of 90 seconds
  esophageal intubation, bleeding, tracheal perforation
Overall success rate | within 48 hours of intubation
  Include all intubation event

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital Zhong-Xing branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Driver B, Dodd K, Klein LR, Buckley R, Robinson A, McGill JW, Reardon RF, Prekker ME. The Bougie and First-Pass Success in the Emergency Department. Ann Emerg Med. 2017 Oct;70(4):473-478.e1. doi: 10.1016/j.annemergmed.2017.04.033. PMID 28601269
- [Background] Ueda W, Arai YP. The Use of a Stylet to Aid the Lifting of the Epiglottis With a Video Laryngoscope. Anesth Pain Med. 2016 May 24;6(4):e38507. doi: 10.5812/aapm.38507. eCollection 2016 Aug. PMID 27843782